CLINICAL TRIAL: NCT05787938
Title: The Role of Magnetic Resonance Imaging in Assessment of the Urinary Bladder Wall Post Transurethral Tumor Resection
Brief Title: Role of MRI in Assessment of the Urinary Bladder Wall Post Transurethral Tumor Resection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Ibrahim Aboelela, Doctor, Assiut University
Other Study IDs: MRI in urinary bladder tumors
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — A procedure that uses radio waves, a powerful magnet, and a computer to make a series of detailed pictures of areas inside the body. A contrast agent, such as gadolinium, may be injected into a vein to help the tissues and organs show up more clearly in the picture. MRI may be used to help diagnose disease, plan treatment, or find out how well treatment is working. It is especially useful for imaging the brain and spinal cord, the heart and blood vessels, the bones, joints, and other soft tissues, the organs in the pelvis and abdomen, and the breast. Also called magnetic resonance imaging, NMRI, and nuclear magnetic resonance imaging.

SUMMARY:
To study the feasibility of using magnetic resonance imaging (MRI) in evaluation UB wall thickening after transurethral resection (TUR) of bladder cancer.

DETAILED DESCRIPTION:
Urinary bladder carcinoma is the second most common tumour of the urinary tract and 70% of such carcinomas are non-muscle-invasive (superficial) at presentation. Transurethral resection (TUR) is the standard treatment; however, recurrence of the tumour is not uncommon so such patients require long-term close supervision.

Staging is based on TNM system. Ta tumors are treated with transurethral resection of bladder tumor (TUR-BT). T1 and carcinoma in situ (Tis) tumors have risk of progression and intravesical immunotherapy with Bacillus-Calmette-Guerin (BCG) instillations is used to obtain local control and organ preservation. Invasive bladder cancer (MIBC) is an aggressive disease and standard treatment is radical cystectomy (RC), accompanied by pelvic lymph node dissection (PLND). In addition to radical surgery, neoadjuvant chemotherapy (NAC) has been demonstrated to increase overall survival in MIBC and is recommended by consensus guidelines.

Compared to contrast enhanced CT, MRI has better soft tissue contrast which may improve local tumor evaluation.

Surveillance strategies for urinary bladder carcinoma recurrence have historically relied on cystoscopy, but this procedure has drawbacks, including its high cost, invasiveness and the fact that it may lead to iatrogenic bladder injury and urinary sepsis. In addition, it cannot diagnose upper tract tumours. The presence of a radiological method that could differentiate between benign and malignant lesions of the bladder would avoid the need for invasive cystoscopy, provided that upper tract tumours were excluded. Diffusion-weighted (DW) MRI is a non-invasive technique measuring the microscopic mobility of water molecules in the tissues without contrast administration. It provides information on perfusion and diffusion simultaneously in any organ, so it can be used to differentiate normal and abnormal structures of tissues, and it might help in the characterization of various abnormalities.

During follow-up of patients after trans-urethral resection (TUR), it is difficult to distinguish residual cancer from fibrotic and inflammatory changes secondary to TUR and intravesical chemotherapy, both of which manifest as bladder wall thickening on T2-weighted MRI.

ELIGIBILITY:
Inclusion Criteria:

-Patients who had a history of TUR of superficial bladder tumors and fit for the MRI examination.

Exclusion Criteria:

* Patients with pacemaker, claustrophobia or metallic prosthesis which are not MRI compatible.
* Patients with contraindications for cystoscopy (unfit for anesthesia or urethral stricture).
* Patients refusing consent for the study.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a history of TUR of superficial bladder tumors. mainly in older people over the age of 55. most common in men, but it's less common in women.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The Role of Magnetic Resonance Imaging (MRI) in assessment of the urinary bladder wall transurethral tumor resection. | Baseline
  To study the feasibility of using magnetic resonance imaging (MRI) in evaluation UB wall thickening after transurethral resection (TUR) of bladder cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Farouk Muorad, Prof.Doctor, Principal Investigator — Assiut University; Mohamed Moamen Elbaroudy, doctor, Principal Investigator — Assiut University

REFERENCES:
- [Background] El-Assmy A, Abou-El-Ghar ME, Refaie HF, Mosbah A, El-Diasty T. Diffusion-weighted magnetic resonance imaging in follow-up of superficial urinary bladder carcinoma after transurethral resection: initial experience. BJU Int. 2012 Dec;110(11 Pt B):E622-7. doi: 10.1111/j.1464-410X.2012.11345.x. Epub 2012 Jul 3. PMID 22757606
- [Background] Wang Y, Zhang W, Xiao W, Chen S, Wei Y, Luo M. Feasibility of Early Evaluation for the Recurrence of Bladder Cancer after Trans-Urethral Resection: A Comparison between Magnetic Resonance Imaging and Multidetector Computed Tomography. Tomography. 2022 Dec 22;9(1):25-35. doi: 10.3390/tomography9010003. PMID 36648990
- [Background] Webb JA. Imaging in haematuria. Clin Radiol. 1997 Mar;52(3):167-71. doi: 10.1016/s0009-9260(97)80269-3. No abstract available. PMID 9091250
- [Background] Le Bihan D, Breton E, Lallemand D, Aubin ML, Vignaud J, Laval-Jeantet M. Separation of diffusion and perfusion in intravoxel incoherent motion MR imaging. Radiology. 1988 Aug;168(2):497-505. doi: 10.1148/radiology.168.2.3393671.
- [Background] Dobson MJ, Carrington BM, Collins CD, Ryder WD, Read G, Hutchinson CE, Hawnaur JM. The assessment of irradiated bladder carcinoma using dynamic contrast-enhanced MR imaging. Clin Radiol. 2001 Feb;56(2):94-8. doi: 10.1053/crad.2000.0560. PMID 11222064